CLINICAL TRIAL: NCT01299558
Title: An Open-label, Non-randomised, Three-way Crossover, Single Dose Study to Determine the Absolute Bioavailability of Fluticasone Furoate (FF)/GW642444 Inhalation Powder, in Healthy Subjects
Brief Title: Study to Look at and Compare How Inhaled and Intravenous Fluticasone Furoate and GW642444 Are Processed by the Body in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 102934
Record Dates: First submitted 2010-06-10; First posted 2011-02-18 (Estimated); Last update posted 2017-06-12 (Actual); Status verified 2017-06

CONDITIONS: Asthma
Keywords: pharmacokinetics; GW642444; absolute bioavailability; healthy subjects; fluticasone furoate; GW685698
MeSH Terms: conditions — Asthma | interventions — fluticasone furoate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Treatment period 1 (Other): Single inhaled dose of FF (800mcg)/GW642444M (100mcg) Inhalation Powder given once daily in the morning on Day 1 of Treatment period 1
  Interventions: Drug: fluticasone furoate//GW642444
- Treatment Period 2 (Other): Single IV dose of FF (250mcg) given over 20 mins on Day 1 of Treatment period 2
  Interventions: Drug: fluticasone furoate
- Treatment Period 3 (Other): Single IV dose of GW642444M (55mcg) given over 60 mins on Day 1 of Treatment period 3
  Interventions: Drug: GW642444

INTERVENTIONS:
Drug: fluticasone furoate//GW642444 — Single inhaled dose of FF (800mcg)/GW642444M (100mcg) Inhalation Powder administered in the morning
  Arms: Treatment period 1
Drug: fluticasone furoate — Single IV dose of FF (250mcg)
  Arms: Treatment Period 2
Drug: GW642444 — Single IV dose of GW642444 (55mcg)
  Arms: Treatment Period 3

SUMMARY:
This study is being done to look at the absolute bioavailability of fluticasone furoate and GW642444 inhalation powder when administered in healthy subjects. Bioavailability is determined by measuring the amount of the dose of inhaled medication that reaches the circulation; the amount of inhaled fluticasone furoate and GW642444 powder will be compared to the medication administered intravenously (where bioavailability is 100%).

DETAILED DESCRIPTION:
Fluticasone furoate (FF), a novel glucocorticoid, and GW642444, a potent, inhaled longacting, beta2-receptor agonist (LABA), are currently under development in combination for use as a once-daily, inhaled treatment for asthma and chronic obstructive pulmonary disease (COPD). FF is also being developed as a stand-alone product for asthma and GW642444 is also being developed as a stand-alone product and in combination with a novel, long-acting muscarinic antagonist for the treatment of COPD. This study is being performed to determine the absolute bioavailability of both FF and GW642444 when delivered in combination from the novel dry powder inhaler.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female between 18 and 64 years of age inclusive
* Body mass index (BMI) within the range 18.5-29 0 kg/m2 (inclusive)
* Subjects who are current non-smokers
* AST, ALT, alkaline phosphatase and bilirubin ≤ 1.5xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%)
* QTcF < 450 msec; or QTc < 480 msec in subjects with Bundle Branch Block, based on a single ECG value, or an average from three ECGs obtained over a brief recording period
* No significant abnormality on the Holter ECG at screening
* FEV1 ≥ 85% predicted at screening.
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form
* Subjects who are able to use the inhalation device satisfactorily

Exclusion Criteria:

* As a result of medical interview, physical examination or screening investigations, the principal investigator or delegate physician deems the subject unsuitable for the study. Subjects must not have a systolic blood pressure above 145 mmHg or a diastolic pressure above 85 mmHg
* Any history of breathing problems in adult life
* Pregnant or lactating females
* The subject has been treated for or diagnosed with depression within six months of screening or has a history of significant psychiatric illness
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones)
* Subjects who have suffered a lower respiratory tract infection within 4 weeks of the screening visit
* Subjects with recent history (within 6 months) of pneumonia
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation
* Any adverse reaction including immediate or delayed hypersensitivity to any beta2-agonist, sympathomimetic drug, or any intranasal, inhaled, or systemic corticosteroid therapy. Known or suspected sensitivity to the constituents of the new powder inhaler (i.e., lactose or magnesium stearate)
* History of milk protein allergy
* Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety
* The subject has taken oral corticosteroids less than 8 weeks before the screening visit
* The subject has taken inhaled, intranasal or topical steroids less than 4 weeks before the screening visit
* History of alcohol/drug abuse or dependence within 12 months of the study
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer)
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period
* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening.
* The subject has tested positive for HIV antibodies
* A positive pre-study urine drug screen or when randomly tested during the study
* Positive carbon monoxide (CO) or alcohol breath test at screening or on admission to the Unit.
* Positive urine cotinine test at screening
* Consumption of seville oranges, pomelos (members of the grapefruit family) or grapefruit juice from 7 days prior to the first dose of study medication
* Unwillingness or inability to follow the procedures outlined in the protocol
* Subject is mentally or legally incapacitated

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2010-05-17 (Actual); Primary Completion 2010-07-15 (Actual); Study Completion 2010-07-15 (Actual)

PRIMARY OUTCOMES:
Absolute bioavailability of FF and GW642444 following single dose of FF/GW642444M Inhalation Powder; determined by measuring the amount of the dose of inhaled medication that reaches the circulation compared to the medication administered intravenously | Up to 48hr PK sampling periods profiles on 3 separate occasions over a total period of up to 5 weeks

SECONDARY OUTCOMES:
Pharmacokinetic parameters: AUC, Cmax, t1/2, tmax, and MRT for all treatments. In addition, volume of distribution (V) and plasma clearance (CL) for intravenous administrations and mean absorption time (MAT) for inhaled treatments | Up to 48hr PK sampling periods profiles on 3 separate occasions over a total period of up to 5 weeks
Number of Participants with clinically significant changes to Vital Signs as a measure of Safety and Tolerability | Approximately 9 weeks for each subject
Number of Participants with clinically significant changes to 12-lead ECG Tests as a measure of Safety and Tolerability | Approximately 9 weeks for each subject
Number of Participants with clinically significant changes to Clinical Laboratory Tests as a measure of Safety and Tolerability | Approximately 9 weeks for each subject
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | Approximately 9 weeks for each subject

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Randwick, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Results for study 102934 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/102934?search=study&study_ids=102934#rs
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Statistical Analysis Plan: 102934 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 102934 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 102934 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 102934 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 102934 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 102934 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 102934 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register